CLINICAL TRIAL: NCT03050229
Title: SGLT-2i and ARB Combination Therapy in Patients With T2DM and Nocturnal Hypertension (SACRA Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jichi Medical University (Other)
Collaborators: Boehringer Ingelheim (Industry); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Kazuomi Kario, Professor & Chairman, Division of Cardiovascular Medicine, Department of Medicine, Jichi Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1245-131
Record Dates: First submitted 2016-12-26; First posted 2017-02-10 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Nocturnal Hypertension; T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Empagliflozin (Experimental): Empagliflozin 10mg/day is administrated orally before or after breakfast for 12 weeks while continuing the existing treatment for hypertension (include AngiotensinII Receptor Blocker [ARB]) and diabetes.
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): Placebo is administrated orally before or after breakfast for 12 weeks while continuing the existing treatment for hypertension (include AngiotensinII Receptor Blocker [ARB]) and diabetes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin 10mg/day once daily before or after breakfast
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Placebo — Placebo once daily before or after breakfast
  Arms: Placebo

SUMMARY:
To explore the beneficial effects of 'empagliflozin + ARB' in comparison with 'placebo + ARB' on the reduction of nocturnal blood pressure in T2DM with hypertension

DETAILED DESCRIPTION:
The study consists of a 8-week run-in period and a 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the following criteria at the start of treatment are eligible for the study:

* Receiving stable treatment with anti-hypertensive including ARB for at least 8 weeks at baseline (0W).
* Receiving stable anti-diabetic treatment with/without anti-diabetics for at least 8 weeks at baseline (0W).
* HbA1c>=6.0%, <10%
* Seated office SBP 130-159mmHg or DBP 80-99mmHg
* Nocturnal hypertension (SBP>=115 mmHg) as measured by Home BP during 5days before baseline (0W).
* Age>=20

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for the study:

* History of hypersensitivity to empagliflozin
* Breast-feeding, pregnant, possibly pregnant, or plan to become pregnant
* Treated with insulin or SU
* With renal dysfunction (eGFR<45mL/min/1.73m2)
* With liver dysfunction (AST or ALT is 3 times higher than reference value)
* Hypotension (systolic blood pressure < 90 mmHg)
* With pituitary gland dysfunction or adrenal gland dysfunction
* Heart failure patients whose NYHA class is IV
* Deemed ineligible for the study due to another reason by investigator
* History of diabetic ketoacidosis or diabetic come within 3 months before enrollment
* History of Acute myocardial infarction, unstable angina, cerebrovascular disease, or transient ischemic attack within 3 months before enrollment
* Patients who have undergone percutaneous transluminal coronary angioplasty (PCI) or coronary artery bypass graftin (CABG) within 3 months before enrollment
* Patients received SGLT2 inhibitor within 8 weeks before enrollment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Reduction of nocturnal blood pressure measured by ABPM | 12 weeks

SECONDARY OUTCOMES:
Reduction of Blood pressure measured by ABPM -24h Blood Pressure | 12 weeks
Reduction of Blood pressure measured by ABPM -Daytime Blood Pressure | 12 weeks
Reduction of Blood pressure measured by ABPM -Minimum nocturnal Blood Pressure | 12 weeks
Reduction of Blood pressure measured by ABPM -Nocturnal blood pressure variability | 12 weeks
Reduction of Metabolism-related factors -HbA1c | 12 weeks
Reduction of Metabolism-related factors -body weight | 12 weeks
Reduction of Metabolism-related factors -BMI | 12 weeks
Reduction of Metabolism-related factors -lipids | 12 weeks
Reduction of Metabolism-related factors -uric acid | 12 weeks
Reduction of Metabolism-related factors -HOMA-R | 12 weeks
Reduction of Metabolism-related factors -HOMA-beta | 12 weeks
Change in Sleep efficacy -Sleep scale (Athens insomnia scale) | 12 weeks
Change in Sleep efficacy -Frequency of nocturnal awakening | 12 weeks
Change in Sleep efficacy -Frequency of nocturia | 12 weeks
Changes in the measures of circulating volume -Plasma NT-proBNP | 12 weeks
Changes in the measures of circulating volume -ANP | 12 weeks
Changes in the measures of organ damage -Urinary albumin/creatinine excretion ratio | 12 weeks
Changes in the measures of organ damage -Urinary Na/K | 12 weeks
Changes in the measures of organ damage -eGFR | 12 weeks
Changes in the measures of organ damage -cystatinC | 12 weeks
The correlation between blood pressure and blood glucose control | 12 weeks
The correlation between blood pressure and body weight | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kazuomi Kario, MD, Principal Investigator — Jichi Medical University
Locations (12):
- Japan (12):
  - Fukuoka University Chikushi Hospital, Fukuoka
  - Kotake Hospital, Fukuoka
  - Onga Hospital, Fukuoka
  - Ishiguro Clinic, Gifu
  - Higashiagatsuma-machi National Health Insurance Clinic, Gunma
  - Katsuya Iin, Hyōgo
  - Minamisanriku Hospital, Miyagi
  - Shibuya Clinic, Saitama
  - International University of Health and Welfare Hospital, Tochigi
  - Jichi Medical University hospital, Tochigi
  - Utsunomiya higashi hospital, Tochigi
  - Kato Clinic, Tokyo

REFERENCES:
- [Derived] Kario K, Okada K, Kato M, Nishizawa M, Yoshida T, Asano T, Uchiyama K, Niijima Y, Katsuya T, Urata H, Osuga JI, Fujiwara T, Yamazaki S, Tomitani N, Kanegae H. Twenty-Four-Hour Blood Pressure-Lowering Effect of a Sodium-Glucose Cotransporter 2 Inhibitor in Patients With Diabetes and Uncontrolled Nocturnal Hypertension: Results From the Randomized, Placebo-Controlled SACRA Study. Circulation. 2019 Apr 30;139(18):2089-2097. doi: 10.1161/CIRCULATIONAHA.118.037076. Epub 2018 Nov 29. PMID 30586745